CLINICAL TRIAL: NCT06345755
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, First-in-human Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of VX-407 in Healthy Subjects
Brief Title: A Phase 1 Study to Evaluate Safety, Tolerability, and Pharmacokinetics of VX-407 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX23-407-001
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: Single Ascending Dose (SAD) (Experimental): Participants will be randomized to receive a single dose of different dose levels of VX-407.
  Interventions: Drug: VX-407
- Part A: Placebo (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-407.
  Interventions: Drug: Placebo
- Part B: Multiple Ascending Dose (MAD) (Experimental): Participants will be randomized to receive multiple doses of different dose levels of VX-407. The dose levels will be determined based on the data from Part A.
  Interventions: Drug: VX-407
- Part B: Placebo (Placebo Comparator): Participants will be randomized to receive multiple doses of placebo matched to VX-407.
  Interventions: Drug: Placebo
- Part C: Drug-Drug Interaction (Experimental): Participants will be administered Midazolam (MDZ) in the presence or absence of VX-407. The dose levels will be determined based on the data from Part B.
  Interventions: Drug: VX-407; Drug: Midazolam
- Part D (Experimental): Participants will be randomized to receive VX-407 in 1 of 3 treatment sequences with 3 dosing periods to assess the relative bioavailability of VX-407 formulations and the effect of food on the pharmacokinetics of VX-407.
  Interventions: Drug: VX-407

INTERVENTIONS:
Drug: VX-407 — Solution or Suspension for oral administration.
  Arms: Part A: Single Ascending Dose (SAD); Part B: Multiple Ascending Dose (MAD); Part C: Drug-Drug Interaction
Drug: Placebo — Solution or Suspension for oral administration.
  Arms: Part A: Placebo; Part B: Placebo
Drug: Midazolam — Syrup for oral administration.
  Arms: Part C: Drug-Drug Interaction
Drug: VX-407 — Suspension or Tablets for oral administration.
  Arms: Part D

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and pharmacokinetic parameters of VX-407 in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (kg/m^2)
* A total body weight of greater than (>) 50 kg
* Nonsmoker or ex-smoker for at least 3 months before screening

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Enrollment up to Day 10
Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Enrollment up to Day 23

SECONDARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of VX-407 | From Day 1 up to Day 6
Part B: Maximum Observed Plasma Concentration (Cmax) of VX-407 | Days 1, 7, and 14
Part A: Area Under the Concentration Versus Time Curve (AUC) of VX-407 | From Day 1 up to Day 6
Part B: Area Under the Concentration Versus Time Curve (AUC) of VX-407 | Days 1, 7, and 14
Part C: Area Under the Concentration Versus Time Curve (AUC) of MDZ in Absence and Presence of VX-407 | On Day 1, and Day 15
Part C: Maximum Observed Plasma Concentration (Cmax) of MDZ in Absence and Presence of VX-407 | On Day 1, and Day 15
Part C: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Enrollment up to Day 24
Part D: Maximum Observed Plasma Concentration (Cmax) of VX-407 Tablet Formulation (test) compared to a Suspension Formulation (reference) Under Fasted Conditions | Days 1, 7, and 13
Part D: Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-407 Under Fasted Conditions | Days 1, 7, and 13
Part D: Maximum Observed Plasma Concentration (Cmax) of VX-407 Tablet Formulation Under Fed versus Fasted State | Days 1, 7, and 13
Part D: Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-407 Tablet Formulation Under Fed versus Fasted State | Days 1, 7, and 13
Part D: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Enrollment up to Day 22

CONTACTS AND LOCATIONS:
Locations (2):
- ICON Lenexa, Lenexa, Kansas, United States
- Altasciences Montreal, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Cortinovis M, Perico N, Remuzzi G. The Need for Novel Therapeutic Directions in Autosomal Dominant Polycystic Kidney Disease Patient Care. Clin J Am Soc Nephrol. 2025 Dec 5. doi: 10.2215/CJN.0000000975. Online ahead of print. PMID 41348481